CLINICAL TRIAL: NCT07405190
Title: A Phase II Study of Ivonescimab as Monotherapy or in Combination With Platinum/Pemetrexed Chemotherapy in Patients With Advanced Non-small Cell Lung Cancer (NSCLC) Harboring Actionable Genomic Alterations (AGAs)
Brief Title: Ivonescimab Alone And With Carboplatin/Pemetrexed For NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Summit Therapeutics (Industry)
Responsible Party: Principal Investigator, Jessica Jiyeong Lin, M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26-015
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Lung Cancer (NSCLC); Lung Cancer Non-Small Cell Cancer (NSCLC); Lung Cancer (Non-Small Cell); Lung Cancer - Non Small Cell; Lung Cancer Non Small Cell; Genomic Alterations
Keywords: NSCLC; AGAs; lung cancer; non-small cell; chemotherapy; ivonescimab
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ivonescimab Monotherapy (Experimental): Patients with advanced/metastatic non-small cell lung cancer harboring actionable genomic alterations with disease progression after prior targeted therapies and chemotherapy will receive ivonescimab monotherapy. Ivonescimab will be administered at the pre-determined dose every 3 weeks on day 1 of each cycle (each cycle is 21 days) until disease progression, unacceptable toxicity, withdrawal of consent, or for up to 24 months, whichever occurs first.
  Interventions: Drug: Ivonescimab
- Ivonescimab plus Carboplatin/Pemetrexed (Experimental): Patients with advanced/metastatic non-small cell lung cancer harboring actionable genomic alterations other than epidermal growth factor receptor mutations with disease progression after prior targeted therapies but no prior chemotherapy will receive ivonescimab, carboplatin, and pemetrexed. Ivonescimab will be administered at the pre-determined dose with the pre-determined doses of carboplatin and pemetrexed on day 1 of the first 4 treatment cycles (each cycle is 21 days) or until disease progression, unacceptable toxicity, or withdrawal of consent, whichever occurs first. Patients who have stable disease or response after the first 4 treatment cycles will continue to receive pre-determined doses of ivonescimab and pemetrexed every 3 weeks until disease progression, unacceptable toxicity, withdrawal of consent, or for up to 24 months, whichever occurs first.
  Interventions: Drug: Ivonescimab; Drug: carboplatin; Drug: pemetrexed

INTERVENTIONS:
Drug: Ivonescimab — Ivonescimab is a specially engineered antibody that can attach to both PD-1 and VEGF-A.
  Other Names: AK112; SMT112
Drug: carboplatin — Carboplatin is a type of chemotherapy drug that contains a special form of platinum.
  Other Names: Paraplatin
  Arms: Ivonescimab plus Carboplatin/Pemetrexed
Drug: pemetrexed — Pemetrexed is a type of chemotherapy drug that works by blocking specific substances, called folates, that cancer cells need to grow and multiply.
  Other Names: Alimta
  Arms: Ivonescimab plus Carboplatin/Pemetrexed

SUMMARY:
The goal of this clinical trial is to assess the efficacy of ivonescimab monotherapy in patients with advanced non-small cell lung cancer harboring actionable genomic alterations who have received prior targeted therapies and chemotherapy. This clinical trial also aims to assess the efficacy of ivonescimab plus carboplatin/pemetrexed chemotherapy in patients with advanced non-small cell lung cancer harboring actionable genomic alterations other than epidermal growth factor receptor mutations who have received prior targeted therapies but no chemotherapy. The main questions it aims to answer are:

* Will ivonescimab alone or together with carboplatin/pemetrexed chemotherapy shrink tumors in the clinical trial's patients?
* Will ivonescimab alone or together with carboplatin/pemetrexed chemotherapy effectively influence if the patients' cancer grows, how long the treatment takes to start working, how long the treatment keeps working after it first starts to help, how long the treatment keeps the cancer from getting worse, and overall survival of patients?
* How many patients receiving ivonescimab alone or together with carboplatin/pemetrexed chemotherapy will experience treatment-emergent, treatment-related, immune-related, and especially interesting side effects? Patients receiving ivonescimab alone will receive an intravenous infusion of ivonescimab every 3 weeks for up to 24 months. Patients receiving ivonescimab together with carboplatin/pemetrexed chemotherapy will receive separate intravenous infusions of ivonescimab, pemetrexed, and carboplatin every 3 weeks for 4 cycles (each cycle is 21 days). These patients will continue to receive infusions of ivonescimab and pemetrexed every 3 weeks for up to 24 total months.

DETAILED DESCRIPTION:
This is a phase II, open-label, two-cohort study designed to determine the efficacy of ivonescimab as monotherapy or in combination with carboplatin/pemetrexed chemotherapy in patients with advanced non-small cell lung cancer harboring actionable genomic alterations who have received prior standard-of-care therapies.

Ivonescimab monotherapy will be evaluated in patients with advanced non-small cell lung cancer with actionable genomic alterations after prior standard-of-care targeted therapies and platinum/pemetrexed chemotherapy. Ivonescimab plus carboplatin/pemetrexed combination regimen will be evaluated in patients with advanced non-small cell lung cancer with non-epidermal growth factor receptor actionable genomic alterations after prior standard-of-care targeted therapies (and no prior chemotherapy).

The U.S. Food and Drug Administration has not approved ivonescimab as a treatment for any disease. The U.S. Food and Drug Administration has approved carboplatin and pemetrexed as a treatment option for non-small cell lung cancer harboring actionable genomic alterations.

Ivonescimab, also known as AK112 and SMT112 during development, is a specially engineered antibody that can attach to both PD-1 and VEGF-A. PD-1 is a protein found on immune cells that "turn off" the immune response. VEGF-A is a protein that helps tumors grow new blood vessels. By binding to both proteins, ivonescimab can reactivate immune cells so they can attack the tumor, block blood vessel growth that feeds the tumor, and reduce the tumor's ability to suppress the immune system, making it easier for immune cells to reach and fight the cancer. Carboplatin is a type of chemotherapy drug that contains a special form of platinum. The drug damages DNA inside cancer cells by creating links or bonds between different parts of the DNA that makes it harder for the cancer cells to grow and divide, eventually leading to cell death. Carboplatin works at any stage of the cell's life cycle, not just when the cell is dividing. Carboplatin is currently sold as Paraplatin. Pemetrexed is a type of chemotherapy drug that works by blocking specific substances, called folates, that cancer cells need to grow and multiply. Folates help cells make DNA and other important cell structures. By preventing folates from working, pemetrexed helps slow down or stop the growth of cancer cells. Pemetrexed is currently sold as Alimta.

Patients will receive study treatment for up to 24 months as long as their disease does not progress, treatment does not cause worsening symptoms, they do not have unacceptable side effects, until they demonstrate an inability or unwillingness to receive the medication regimen and/or follow the document requirements, or they withdraw from the study. Patients will be followed for up to 2 years after the last patient is enrolled. It is expected that about 46 people will take part in this research study.

Summit Therapeutics, Inc. is supporting this research study by providing the study drug, ivonescimab, and funding for the clinical trial activities.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced or metastatic non-squamous NSCLC not amenable to curative resection or radiation.
* AGA requirements as follows:

Ivonescimab monotherapy: Tumor harboring classical EGFR sensitizing mutation (i.e., L858R, exon 19 deletion), or ALK, ROS1, RET, or NTRK1-3 fusion, per local testing. Note: The number of patients with EGFR mutation-positive NSCLC enrolled will be capped at maximum of 10 (in order to ensure the assessment of non-EGFR disease subsets). Ivonescimab plus carboplatin/pemetrexed: Tumor harboring ALK, ROS1, RET, or NTRK1-3 fusion, per local testing.

* Prior therapy requirements as follows:

  a. Prior genotype-specific standard-of-care targeted therapy must have included at least one genotype-appropriate TKI(s) specified below: i. EGFR sensitizing mutation: a third-generation EGFR TKI such as osimertinib or lazertinib ii. ALK fusion: a third- or fourth-generation ALK TKI such as lorlatinib or neladalkib (NVL-655) iii. ROS1 fusion: crizotinib, entrectinib, repotrectinib, or taletrectinib iv. RET fusion: selpercatinib or pralsetinib v. NTRK1-3 fusion: entrectinib, larotrectinib, or repotrectinib Ivonescimab monotherapy: Must have received platinum/pemetrexed chemotherapy. No limitations on the number of prior lines of systemic therapy including the number of lines of chemotherapy or TKI(s). Ivonescimab plus carboplatin/pemetrexed: May not have received any prior chemotherapy. No limitations on the number of prior TKI(s).
* At least 1 measurable lesion as assessed by investigator per the RECIST v1.1 criteria for both cohorts.
* Participants must be willing to undergo the mandatory pre-treatment and post-progression tissue biopsies. If archival pre-treatment tissue is available from within 6 months of study enrollment, with no new intervening systemic therapy since the biopsy, a repeat pre-treatment biopsy may be omitted upon discussion with the principal investigator. On-treatment tissue biopsy (obtained within 7 days prior to Cycle 2 Day 1) will be mandatory for patients in Cohort 1 and optional for patients in Cohort 2. In select cases, if medically deemed unsafe/not feasible, exception may be granted upon discussion with the principal investigator.
* Clinically asymptomatic treated or untreated brain metastases are allowed if they have not required increasing doses of steroids within 2 weeks prior to study entry for CNS symptoms.
* Age ≥18 years old.
* ECOG performance status of 0 or 1.
* Adequate Organ Function:

  a. Hematology (no blood transfusions or growth factor therapy used within 7 days of the screening CBC): i. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L ii. Platelet count ≥ 100 × 109/L iii. Hemoglobin ≥ 9.0 g/dL b. Kidneys: i. Creatinine clearance (CrCl) ≥ 50 mL/min using the Cockcroft-Gault formula (Cohorts 1 and 2) or estimated glomerular filtration rate (eGFR) value ≥ 60 mL/min (for Cohort 1) or ≥30 mL/min (for Cohort 2) using the Cockcroft-Gault formula or estimated glomerular filtration rate (eGFR) ii. Urine protein < 2+ or 24 hour urine protein quantification < 1.0 g c. Liver: i. Serum total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN); for patients with liver metastases or confirmed/suspected Gilbert syndrome, TBIL ≤3 × ULN ii. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT)
  * 2.5 × ULN; for patients with liver metastases, AST and ALT ≤ 5 × ULN d. Coagulation: prothrombin time (PT) or international normalized ratio (INR)
  * 1.5 x ULN, and partial prothrombin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN (unless abnormalities are unrelated to coagulopathy). This applies only to patients who are not on therapeutic anti-coagulation. Patients receiving therapeutic anti-coagulation should be on a stable dose for at least one month prior to study enrollment.
* Female patients of childbearing age must have negative serum pregnancy test results before first ivonescimab drug dose or per region-specific guidance documented in the informed consent and a negative urine pregnancy test on the day of first dose prior to dosing.
* Female patient of childbearing potential having sex with an unsterilized male partner must agree to use a highly effective method of contraception from the beginning of screening until 90 days after the last dose of the ivonescimab and until 6 months after the last doses of carboplatin and pemetrexed.
* Unsterilized male patients having sex with a female partner of childbearing potential, or a pregnant or breastfeeding partner must agree to use barrier contraception (male condom) for the duration of the treatment period until 90 days after the last dose of ivonescimab and until 90 days after the last doses of carboplatin and pemetrexed. Male patients with female partners of childbearing potential must have the female partner agree to use at least 1 form of highly effective contraception for the duration of the treatment period until 90 days after the last dose of ivonescimab and until 90 days after the last doses of carboplatin and pemetrexed.

Exclusion Criteria:

* Participants previously treated with immune checkpoint inhibitors or other T cell immune-modulating antibodies, including anti-CTLA-4, anti-PD-1 and/or anti-PD-L1 agents.
* Major surgical procedures or serious trauma within 4 weeks prior to first ivonescimab dose or plans for major surgical procedures within 4 weeks after the first ivonescimab dose (as determined by the investigator). Minor local procedures (excluding central venous catheterization and port implantation) within 3 days prior to first ivonescimab dose.
* History of bleeding tendencies or coagulopathy and/or clinically significant bleeding symptoms or risk within 4 weeks prior to first ivonescimab dose, including but not limited to:

  1. Hemoptysis (defined as coughing up ≥ 0.5 teaspoon of fresh blood or small blood clots). Note: transient hemoptysis associated with diagnostic bronchoscopy is allowed.
  2. Nasal bleeding/epistaxis (bloody nasal discharge is allowed)
  3. Current use of prophylactic or full-dose anticoagulants or anti-platelet agents for therapeutic purposes that is not stable prior to first ivonescimab dose is not allowed; stability of anti-coagulation dosing will be defined by remaining on the same dose for at least one month prior to study enrollment.
  4. The use of full-dose anticoagulants is permitted as long as the international normalized ratio (INR) or activated partial thromboplastin time (aPTT) is within therapeutic limits according to the medical standard of the enrolling institution.
* Poorly controlled hypertension with repeated systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg after oral antihypertensive therapy.
* Active autoimmune or lung disease requiring systemic therapy (eg, with disease modifying drugs, prednisone >10 mg daily or equivalent, immunosuppressant therapy) within 2 years prior to first ivonescimab dose; however, the following will be allowed:

  1. Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is permitted.
  2. Intermittent use of bronchodilators, inhaled corticosteroids, or local corticosteroid injections is permitted.
* History of major diseases before first ivonescimab dose, specifically:

  1. Unstable angina, myocardial infarction, congestive heart failure (New York Heart Association [NYHA] classification ≥ grade 2) or unstable vascular disease (eg, aortic aneurysm at risk of rupture, Moyamoya disease) that required hospitalization within 6 months prior to first ivonescimab dose, or other cardiac impairment that may affect the safety evaluation of the study drug (eg, poorly controlled arrhythmias, myocardial ischemia)
  2. History of esophageal gastric varices, severe ulcers, wounds that do not heal, abdominal fistula, intra-abdominal abscesses, or acute gastrointestinal bleeding within 6 months before first ivonescimab dose
  3. History of any grade arterial thromboembolic event, Grade 3 and above venous thromboembolic event, as specified in National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 6.0, transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy within 6 months prior to first ivonescimab dose
  4. Acute exacerbation of chronic obstructive pulmonary disease within 4 weeks before first ivonescimab dose
  5. History of perforation of the gastrointestinal tract and/or fistula, history of gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection) within 6 months prior to first ivonescimab dose
* Imaging during the screening period shows that the patient has:

  1. Radiologically documented evidence of major blood vessel invasion (central pulmonary artery, central pulmonary veins, aorta, brachiocephalic artery, common carotid artery, subclavian artery, superior vena cava) or tumor invading organs (heart, trachea, esophagus, central bronchi [not including segmental bronchi]) or if there is a risk of esophagotracheal or esophagopleural fistula in the opinion of the investigator.
  2. Radiographic evidence of major blood vessel encasement with narrowing of the vessel or intratumor lung cavitation or necrosis that the investigator determines will pose a significantly increased risk of bleeding.
* Symptomatic CNS metastases, CNS metastases with hemorrhagic features, CNS metastasis ≥ 1.5 cm, CNS radiation within 7 days prior to first ivonescimab dose, potential need for CNS radiation within the first cycle, or leptomeningeal disease.

Note: Patients must have stopped corticosteroids or be on physiologic corticosteroid replacement therapy (prednisone ≤ 10 mg daily or equivalent).

* Live vaccine or live attenuated vaccine within 4 weeks prior to planned first ivonescimab dose, or if scheduled to receive a live vaccine or live attenuated vaccine during the study period. Inactivated vaccines are permitted.
* Severe infection within 4 weeks prior to first ivonescimab dose, including but not limited to comorbidities requiring hospitalization, sepsis, or severe pneumonia; active infection (as determined by the investigator) requiring systemic anti-infective therapy within 2 weeks prior to first ivonescimab dose (excluding antiviral therapy for hepatitis B or C)
* Has pre-existing peripheral neuropathy that is ≥ Grade 2 by CTCAE version 6
* Uncontrolled pleural effusions, pericardial effusions, or ascites that is clinically symptomatic Note: Patients managed with indwelling catheters (eg, PleurX) are allowed.
* Any evidence of current ILD or pneumonitis or a prior history of ILD or non-infectious pneumonitis requiring systemic corticosteroids
* Active or prior history of inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis, or chronic diarrhea)
* Known history of human immunodeficiency virus (HIV) whose viral load is not controlled.
* Current use of systemic corticosteroids (>10 mg daily prednisone or equivalent)
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation
* Patients with active hepatitis B are required to have stable or declining levels of hepatitis B DNA by polymerase chain reaction (PCR) on appropriate anti-viral therapy with acceptable tolerability for one month prior to first ivonescimab dose. All patients with active hepatitis C (hepatitis C virus [HCV] antibody positive with HCV RNA levels above the lower limit of detection) are excluded.
* Known allergy to any component of any study drug; known history of severe hypersensitivity to other monoclonal antibodies
* History or current evidence of any condition (medical [including adverse events from prior anticancer therapy, disorders secondary to tumor], surgical or psychiatric [including substance abuse]), or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, might lead to higher medical risk and/or is not in the best interest of the patient to participate, in the opinion of the treating investigator
* Patient is breastfeeding or plans to breastfeed during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-08-04 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) of Ivonescimab Monotherapy | Day 1 of cycle 1 (each cycle is 21 days) to disease progression, loss of follow-up, withdrawal of consent, study termination, or for up to 2 years from the day the last patient is enrolled, whichever occurs first.
  The objective response rate (ORR) is defined as the number of patients with confirmed best overall response or complete response or partial response (PR) divided by the number of treated patients in the cohort. ORR will be measured per investigator. BOR will be assessed per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria.
Objective Response Rate (ORR) of Ivonescimab plus Carboplatin/Pemetrexed | Day 1 of cycle 1 (each cycle is 21 days) to disease progression, loss of follow-up, withdrawal of consent, study termination, or for up to 2 years from the day the last patient is enrolled, whichever occurs first.
  The objective response rate (ORR) is defined as the number of patients with confirmed best overall response or complete response or partial response (PR) divided by the number of treated patients in the cohort. ORR will be measured per investigator. BOR will be assessed per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) of Ivonescimab Monotherapy | Day 1 of cycle 1 (each cycle is 21 days) to disease progression, loss of follow-up, withdrawal of consent, study termination, or for up to 2 years from the day the last patient is enrolled, whichever occurs first.
  Disease control rate (DCR) is defined as the percentage of participants who have either a complete response, partial response, or stable disease. DCR will be assessed per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria.
Disease Control Rate (DCR) of Ivonescimab plus Carboplatin/Pemetrexed | Day 1 of cycle 1 (each cycle is 21 days) to disease progression, loss of follow-up, withdrawal of consent, study termination, or for up to 2 years from the day the last patient is enrolled, whichever occurs first.
  Disease control rate (DCR) is defined as the percentage of participants who have either a complete response, partial response, or stable disease. DCR will be assessed per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria.
Time to Response (TTR) of Ivonescimab Monotherapy | Day 1 of cycle 1 (each cycle is 21 days) to the first documentation of complete or partial response for up to 2 years from the day the last patient is enrolled.
  Time to response (TTR) is defined as the amount of time between the first dose of ivonescimab to the first time that measurement criteria are met for complete response or partial response. TTR will be assessed per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria.
Time to Response (TRR) of Ivonescimab plus Carboplatin/Pemetrexed | Day 1 of cycle 1 (each cycle is 21 days) to the first documentation of complete or partial response for up to 2 years from the day the last patient is enrolled.
  Time to response (TTR) is defined as the amount of time between the first doses of ivonescimab, carboplatin, and pemtrexed to the first time that measurement criteria are met for complete response or partial response. TTR will be assessed per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria.
Duration of Response (DOR) of Ivonescimab Monotherapy | First day complete or partial response is recorded to the first day progressive disease is recorded or, if no progressive disease occurs, the date of last radiological assessment up to 2 years from the day the last patient is enrolled.
  Duration of response (DOR) is defined as the amount of time from the first recording of complete or partial response (whichever is recorded first) to the first date that progressive disease is objectively documented. DOR will be assessed per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria. Patients who do not achieve at least a partial response, will be excluded from the analysis of DOR.
Duration of Response (DOR) of Ivonescimab plus Carboplatin/Pemetrexed | First day complete or partial response is recorded to the first day progressive disease is recorded or, if no progressive disease occurs, the date of last radiological assessment up to 2 years from the day the last patient is enrolled.
  Duration of response (DOR) is defined as the amount of time from the first recording of complete or partial response (whichever is recorded first) to the first date that progressive disease is objectively documented. DOR will be assessed per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria. Patients who do not achieve at least a partial response, will be excluded from the analysis of DOR.
Progression-Free Survival (PFS) of Ivonescimab Monotherapy | Day 1 of cycle 1 (each cycle is 21 days) to the first day of documented disease progression, death, or if no disease progression or death occurs, the day of the last radiological assessment, up to 2 years from the day the last patient was enrolled.
  Progression-free survival (PFS) is defined as the time from the start date of the study drug treatment to the date of first documented progression or death due to any cause. PFS will be assessed will be assessed per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria. PFS will be summarized using the Kaplan-Meier method with median PFS time (including two-sided 95% confidence interval (CI)). The PFS rates at 6 months and at 12 months will be estimated with two-sided 95% CIs.
Progression-Free Survival (PFS) of Ivonescimab plus Carboplatin/Pemetrexed | Day 1 of cycle 1 (each cycle is 21 days) to the first day of documented disease progression, death, or if no disease progression or death occurs, the day of the last radiological assessment, up to 2 years from the day the last patient was enrolled.
  Progression-free survival (PFS) is defined as the time from the start date of the study drug treatment to the date of first documented progression or death due to any cause. PFS will be assessed will be assessed per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria. PFS will be summarized using the Kaplan-Meier method with median PFS time (including two-sided 95% confidence interval (CI)). The PFS rates at 6 months and at 12 months will be estimated with two-sided 95% CIs.
Overall Survival (OS) of Ivonescimab Monotherapy | Day 1 of cycle 1 (each cycle is 21 days) to death, day of last consent for patients who are lost to follow-up or withdraw, or the study cutoff date for patients will receiving treatment, up to 2 years from the day the last patient was enrolled.
  Overall survival (OS) is defined as the time from the start date of the study drug treatment to death due to any cause. OS will be assessed will be assessed per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria. OS will be summarized using the Kaplan-Meier method with median OS time (including two-side 95% confidence interval (CI)). The OS rates at 6, 12, 18, and 24 months will be estimated with two-sided 95% CIs.
Overall Survival (OS) of Ivonescimab plus Carboplatin/Pemetrexed | Day 1 of cycle 1 (each cycle is 21 days) to death, day of last consent for patients who are lost to follow-up or withdraw, or the study cutoff date for patients will receiving treatment, up to 2 years from the day the last patient was enrolled.
  Overall survival (OS) is defined as the time from the start date of the study drug treatment to death due to any cause. OS will be assessed will be assessed per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria. OS will be summarized using the Kaplan-Meier method with median OS time (including two-side 95% confidence interval (CI)). The OS rates at 6, 12, 18, and 24 months will be estimated with two-sided 95% CIs.
Number of Patients who Experience Adverse Events and Serious Adverse Events on Ivonescimab Monotherapy | Day 1 of cycle 1 (each cycle is 21 days) to the day 90 follow-up visit.
  The number of patients with treatment-emergent and treatment-related adverse events (AEs) and serious AEs (SAEs) will be assessed by Common Terminology Criteria for Adverse Events (CTCAE) v6.0. The number and percentage of participants who experience any AE, SAE, treatment-related AE, and treatment-related SAE will be summarized according to worst toxicity grades.
Number of Patients who Experience Adverse Events and Serious Adverse Events on Ivonescimab plus Carboplatin/Pemetrexed | Day 1 of cycle 1 (each cycle is 21 days) to the day 90 follow-up visit.
  The number of patients with treatment-emergent and treatment-related adverse events (AEs) and serious AEs (SAEs) will be assessed by Common Terminology Criteria for Adverse Events (CTCAE) v6.0. The number and percentage of participants who experience any AE, SAE, treatment-related AE, and treatment-related SAE will be summarized according to worst toxicity grades.
Number of Patients who Experience Immune-Related and Especially Interesting Adverse Events on Ivonescimab Monotherapy | Day 1 of cycle 1 (each cycle is 21 days) to the 90 day follow-up visit.
  Frequency, management, and resolution of select immune-related adverse events (irAEs) and adverse events of special interest (AESIs) will be analyzed. Time-to onset, severity, duration of irAEs and AESIs, action taken with the study drug, dosing delays, corticosteroid details, and re-challenge information will be recorded.
Number of Patients who Experience Immune-Related and Especially Interesting Adverse Events on Ivonescimab plus Carboplatin/Pemetrexed | Day 1 of cycle 1 (each cycle is 21 days) to the 90 day follow-up visit.
  Frequency, management, and resolution of select immune-related adverse events (irAEs) and adverse events of special interest (AESIs) will be analyzed. Time-to onset, severity, duration of irAEs and AESIs, action taken with the study drug, dosing delays, corticosteroid details, and re-challenge information will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jessics J Lin, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: Jessica Lin, MD at 617-724-4000 or jjlin1@partners.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovation team at http://www.partners.org/innovation